CLINICAL TRIAL: NCT01653860
Title: Partner Violence and Anger Management: a Randomised Controlled Study of the Effectiveness of Cognitive Behavioral Therapy
Brief Title: Partner Violence and Anger Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012/683
Record Dates: First submitted 2012-07-25; First posted 2012-07-31 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Domestic Violence; Spouse Abuse
Keywords: Behavior therapy; Group therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Brøset anger management model (Experimental): Group treatment
  Interventions: Behavioral: The Brøset anger management model
- ordinary group treatment (Active Comparator): Group treatment
  Interventions: Behavioral: Ordinary group treatment

INTERVENTIONS:
Behavioral: The Brøset anger management model — manualised structured cognitive treatment program 15 weeks (30 hours)
  Arms: The Brøset anger management model
Behavioral: Ordinary group treatment — group treatment 8 weeks (16 hours)
  Arms: ordinary group treatment

SUMMARY:
The purpose of this study is to investigate the effectiveness of the Brøset anger management model in reducing violent behavior amongst clients who are violent in intimate partnerships and who voluntarily seek help.

Violence in intimate partnerships constitutes a serious problem worldwide and there is reason to believe that cognitive behavior therapy has some effect on the reduction of violent behavior. However, there are currently too few randomized controlled studies to conclude about the effectiveness of cognitive behavior therapy for this client group.

ELIGIBILITY:
Inclusion Criteria:

* fluent in Norwegian language
* is in a partner relationship at inclusion. Partner relationship is defined by having an intimate partner at present, or being in regular contact with a former intimate partner so that violence is possible (e.g. they have children)
* admits being violent to his partner (physical, mental and/or sexual)

Exclusion Criteria:

* psychosis
* alcohol- or drug addiction to a level that hinders group participation free from intoxication.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
violent behaviour, reported by partner and client | 3 months between assessments, 1 year duration, i.e. baseline and 4 follow-up assessments. In accordance with the original Norwegian protocol.
  measured by using the Conflict Tactics Scale Revised (CTS2), instrument for measuring violence in intimate partnerships(10), which consists of 78 questions (0-7) about different aspects of violence (frequence of physical, psychological, sexual and material violence)

SECONDARY OUTCOMES:
The client's and their partner's mental health | 3 months between assessments, 1 year duration, i.e. baseline and 4 follow-up assessments. In accordance with the original Norwegian protocol.
  measured by using the Hopkins Symptoms Check List (HSCL-25, with 25 questions about the presence and intensity of anxiety and depression symptoms, and symptoms of somatoform character)
The client's and their partner's health service use and absence due to sickness | 3 months between assessments, 1 year duration, i.e. baseline and 4 follow-up assessments. In accordance with the original Norwegian protocol.
Changes in emotional dysregulation | 3 months between assessments, 1 year duration, i.e. baseline and 4 follow-up assessments. In accordance with the original Norwegian protocol.
  Emotional regulation will be assessed by the Difficulties in Emotion Regulation Scale (DERS, Gratz & Roemer, 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Tom Palmstierna, MD PhD prof, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St Olavs University Hospital, Division of Psychiatry, Centre for research and education in forensic psychiatry Brøset, Trondheim, Norway

REFERENCES:
- [Result] Nesset MB, Lara-Cabrera ML, Bjorngaard JH, Whittington R, Palmstierna T. Cognitive behavioural group therapy versus mindfulness-based stress reduction group therapy for intimate partner violence: a randomized controlled trial. BMC Psychiatry. 2020 Apr 19;20(1):178. doi: 10.1186/s12888-020-02582-4. PMID 32306935
- [Result] Nesset MB, Bjorngaard JH, Whittington R, Palmstierna T. Does cognitive behavioural therapy or mindfulness-based therapy improve mental health and emotion regulation among men who perpetrate intimate partner violence? A randomised controlled trial. Int J Nurs Stud. 2021 Jan;113:103795. doi: 10.1016/j.ijnurstu.2020.103795. Epub 2020 Oct 14. PMID 33120137